CLINICAL TRIAL: NCT02332876
Title: Physical Activity and Neuropsychological Outcomes in a Cancer Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 1K07CA181323-01A1 (NIH)
Record Dates: First submitted 2014-12-23; First posted 2015-01-07 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Cognitive Dysfunction; Breast Cancer Survivors
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention (Experimental): This arm will receive a 12-week individually tailored phone and email-based exercise program.
  Interventions: Behavioral: Exercise
- Wellness Waitlist Control (Active Comparator): This arm will receive emails on the same schedule as the exercise arm, that cover a variety of health and wellness topics. At the end of the 12 weeks, participants will be able to start the exercise program.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise Intervention
Behavioral: Control
  Arms: Wellness Waitlist Control

SUMMARY:
Many cancer survivors experience treatment-related impairments in mental abilities such as memory, attention, and concentration (known as cognition). Research indicates that physical activity can improve cognition in healthy adults; however, little is known about whether physical activity can improve cognition among cancer survivors. This study will test whether a physical activity intervention results in improvements in cognition among breast cancer survivors, which may lead to interventions to improve cognition.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer survivors; diagnosed at stage 1, 2, or 3 less than 5 years ago -
* not scheduled for or currently undergoing chemotherapy; sedentary, defined as engaging in less than 60 minutes of moderate to vigorous physical activity each week
* accessible geographically and by telephone
* have access to the internet
* endorse experience difficulties with thinking abilities
* in addition, participants on adjuvant therapy (e.g., tamoxifen or aromatase inhibitors) must be able and willing to remain on that treatment for the 3-month intervention period to prevent confounding of biomarker concentrations by treatment.

Exclusion Criteria:

* history of coronary heart disease, diabetes, stroke, orthopedic conditions that limit mobility, or any other serious medical condition that could make it potentially unsafe to be in an unsupervised physical activity intervention
* other primary or recurrent invasive cancer within the last 10 years (other than nonmelanoma skin cancer or carcinoma of the cervix in situ)
* unable to commit to a 3-month intervention schedule; any condition that, in the investigators' judgment, would contraindicate increased physical activity or otherwise interfere with participation in the trial
* unable to provide a blood sample at the baseline measurement visit
* unable to speak and read English.

Ages: 21 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Hartman SJ, Chen R, Tam RM, Narayan HK, Natarajan L, Liu L. Fitbit Use and Activity Levels From Intervention to 2 Years After: Secondary Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jun 30;10(6):e37086. doi: 10.2196/37086. PMID 35771607
- [Derived] Hartman SJ, Weiner LS, Nelson SH, Natarajan L, Patterson RE, Palmer BW, Parker BA, Sears DD. Mediators of a Physical Activity Intervention on Cognition in Breast Cancer Survivors: Evidence From a Randomized Controlled Trial. JMIR Cancer. 2019 Oct 11;5(2):e13150. doi: 10.2196/13150. PMID 31605514
- [Derived] Weiner LS, Takemoto M, Godbole S, Nelson SH, Natarajan L, Sears DD, Hartman SJ. Breast cancer survivors reduce accelerometer-measured sedentary time in an exercise intervention. J Cancer Surviv. 2019 Jun;13(3):468-476. doi: 10.1007/s11764-019-00768-8. Epub 2019 May 29. PMID 31144265
- [Derived] Hartman SJ, Nelson SH, Weiner LS. Patterns of Fitbit Use and Activity Levels Throughout a Physical Activity Intervention: Exploratory Analysis from a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Feb 5;6(2):e29. doi: 10.2196/mhealth.8503. PMID 29402761

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Intervention: This arm received a Fitbit along with a 12-week individually tailored phone and email-based exercise program.
  Exercise
- Wellness Waitlist Control: This arm will receive emails on the same schedule as the exercise arm, that cover a variety of health and wellness topics. At the end of the 12 weeks, participants will be able to start the exercise program.
  Control
Period: Overall Study
Arm/Group | Exercise Intervention | Wellness Waitlist Control
Started | 43 | 44
Completed | 42 | 43
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention | Wellness Waitlist Control | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.37) | 56.2 (9.30) | 57.2 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 35 | 37 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 1 | 2
  White | 36 | 35 | 71
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health Toolbox - Cognition Domain- Oral Symbol Digit Test
Description: Change in score on the NIH Toolbox Oral Symbol Digit test, an objective measure of processing speed, from baseline to 12 weeks. The Oral Symbol Digit test provides a raw score (possible range is 0-144). A higher score indicates better processing speed.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention | Wellness Waitlist Control
Number analyzed (Participants) | 43 | 44
units on a scale | 7 (10.2) | 3 (8.2)
Statistical Analysis 1: Comparison: Exercise Intervention vs Wellness Waitlist Control; Test type: Superiority; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Exercise Intervention: This arm will receive a 12-week individually tailored phone and email-based exercise program.
  Exercise
Arm/Group | Exercise Intervention | Wellness Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No